CLINICAL TRIAL: NCT00917982
Title: The Effect of Vision Therapy/Orthoptic on Motor & Sensory Status of the 3 to 7
Brief Title: The Effect of Vision Therapy/Orthoptic on Motor & Sensory Status of the 3 to 7 Years Old Strabismic Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Other Study IDs: 8801
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus

ARMS (1):
- Vision therapy (Other)
  Interventions: Other: vision therapy

INTERVENTIONS:
Other: vision therapy

SUMMARY:
Vision therapy (VTO) is a group of non-surgical treatment helping patients in 3 subjects;1)increasing the the visual acuity 2)improving the mechanical skills resulting in increasing the power of extraocular muscles,biocular vision,peripheral vision 3) increasing the perceptual skills making the brain to percept the colour and visual memory better.In this study we are going to compare the effect of vision therapy /orthoptic on motor & sensory of the 3 to 7 years old strabismic patients

ELIGIBILITY:
Inclusion Criteria:

* 3<age<7
* Congenital isotropia

Exclusion Criteria:

* Muscular disease
* General ocular and systemic disease
* Seizure
* Visual Acuity < 60/20
* Nystagmus
* Follow up less than 3 months after surgery

Ages: 3 Years to 7 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran